CLINICAL TRIAL: NCT05587231
Title: Comparison of the Postoperative Use of Dextenza (Dexamethasome Ophthalmic Insert) vs a Standard Regimen of Topical Fluorometholone After PRK
Brief Title: Comparison of the Postoperative Use of Dextenza vs a Standard Regimen After PRK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Navy Medical Center San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2021.0059
Record Dates: First submitted 2022-09-30; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Steroid Ophthalmic Insert
Keywords: Refractive surgery; PRK (photorefractive keratectomy); Dextenza; Fluorometholone
MeSH Terms: interventions — Calcium Dobesilate; Fluorometholone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dextenza 0.4Mg Ophthalmic Insert (Experimental): Dextenza (a dexamethasone ophthalmic insert manufactured by Ocular Therapeutix) will be inserted immediately after PRK surgery to administer a post surgery steroid regimen. No steroid drops will be adminstered.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Topical Fluorometholone (Active Comparator): Standard of care topical Fluorometholone drops will be used by the subjects after PRK Surgery. There will be a taper as follows:
  i. 1 drop in each eye QID for 1st week postop. ii. 1 drop in each eye TID for 2nd week postop. iii. 1 drop in each eye BID for 3rd week postop. iv. 1 drop in each eye qD for 4th week postop.
  Interventions: Drug: Topical Fluorometholone

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — The experimental group will have the Dextenza Insert implanted immediately after surgery
  Arms: Dextenza 0.4Mg Ophthalmic Insert
Drug: Topical Fluorometholone — Steroid drops will be administered by the subject according to the standard of care taper
  Arms: Topical Fluorometholone

SUMMARY:
Naval Refractive Surgery Center proposes a prospective, single-site, randomized, non-FDA regulated clinical trial with bilateral commercial treatment for for PRK. Subjects will be randomized to receive one of two postoperative steroid regimens: Dextenza (a dexamethasone ophthalmic insert) or standard of care topical Fluorometholone. Subjects will be followed for 3 months after surgery. Investigators will use objective and subjective measures to assess potential differences in postoperative healing and pain.

This study will not be FDA-regulated. All study surgeries will be standard of care, with the exception of the addition of the Dextenza insert after the PRK procedure among subjects randomized to the Dextenza group.

DETAILED DESCRIPTION:
The Dextenza in the DoD study is a prospective, randomized, comparative, single-site, non-FDA regulated clinical trial to compare two different postoperative steroid regimens in active duty populations that are treated with PRK at the Navy Refractive Surgery Center in San Diego,California.

Study subjects will be randomly assigned to receive one of two post-PRK steroid regimens:

1. Dextenza (a dexamethasone ophthalmic insert manufactured by Ocular Therapeutix)
2. Standard of care topical Fluorometholone

For each study subject, both eyes will be randomized to the same postoperative steroid regimen. That is, this is a bilateral eye study (not contralateral).

The myopic treatments will range from 0.00 D to -8.00 D MRSE, with cylinder from -0.00 to - 3.00 D (myopia with or without astigmatism). This treatment range is within FDA-approved limits for PRK, as well as all proposed study lasers.

The primary objective of this clinical trial is to evaluate the potential postoperative differences in pain and epithelial closure in active duty subjects treated with PRK at the Navy Refractive Surgery Center. Study subjects will be randomly assigned to receive one of two post-PRK steroid regimens:

1. Dextenza

   1. Dextenza is a 0.4mg dexamethasone ophthalmic insert manufactured by Ocular Therapeutix.
   2. It is placed into the lower lacrimal punctum immediately after PRK (bilaterally).
   3. The insert slowly dissolves over time.
2. Standard of care topical Fluorometholone (0.1% ophthalmic suspension) a. Tapered over time: i. 1 drop in each eye QID for 1 st week postop. ii. 1 drop in each eye TID for 2 nd week postop. iii. 1 drop in each eye BID for 3 rd week postop. iv. 1 drop in each eye qD for 4 th week postop.

This clinical trial is not regulated by the FDA.

The Investiators hypothesize that there will be no statistically significant nor clinically meaningful differences in postoperative self-reported pain or epithelial closure when comparing Dextenza to Fluorometholone. The Investigators also hypothesize that adherence to the medication regimen will be higher in the Dextenza group because it is an ophthalmic insert rather than a topical medication.

These potential differences will be evaluated using the following statistical methods:

Chi-Square tests of dichotomous and categorical Visual Analogue Scale and COMTOL questionnaire responses (within a single time period) between Dextenza and Fluorometholone groups. McNemar's or Marginal Homoegenity tests of categorical Visual Analogue Scale and COMTOL questionnaire responses being compared over study visits between Dextenza and Fluorometholone groups. The Investigators will adjust for multiple comparisons using Bonferroni, Tukey, or Scheffe's methods for adjustment.

This study will be performed in an active duty population. Subjects will undergo Wavefront Guided (VISX or similar) or Wavefront Optimized PRK (e.g., Wavelight EX500 or similar) fr the reduction or elimination of myopia with or without astigmatism.

The following outcomes will include a binocular/subject-level analysis:

-UCVA OU, BSCVA OU, Manifest refraction OU, Subject history, Cycloplegic refraction OU, Intraoperative events, Adverse events, Combat Driving Performance Test, Take Home questionnaire, COMTOL questionnaire, PROWL questionnaire.

The following outcomes will include an analysis of each eye treated independently:

UCVA OD & OS, BSCVA OD & OS, Manifest refraction OD & OS, Cycloplegic refraction OD & OS, Topography, including keratometry OD & OS, Wavefront OD & OS, Dilated fundus exams OD & OS, Pachymetry OD & OS, Slit lamp examinations OD & OS, Intraocular pressure OD & OS, Intraoperative events, Adverse events.

The Navy is uniquely positioned to perform this comparison due to the availability of the study lasers at NMCSD and of a large subject pool and a history of good follow-up in the active duty population.

RANDOMIZATION

1. Subjects will be randomized to receive either receive one of two postoperative steroid regimens:

   * 1) Dextenza insert
   * 2) Topical Fluorometholone regimen
2. Randomization lists will be stratified by preoperative manifest sphere to ensure balanced randomization by refractive error:

   * Low (-1.00 to -3.00 D SPH)
   * Moderate (-3.25 to -6.00 D SPH)
   * High (Greater than -6.00 D SPH)

In cases where each eye falls into a different sphere stratum, the eye with the highest manifest sphere will be used to randomize both of the subject's eyes.

STEROID REGIMEN

Subjects will follow one of two randomly assigned postoperative steroid regimens:

1. Dextenza

   1. Dextenza is a 0.4mg dexamethasone ophthalmic insert manufactured by Ocular Therapeutix.
   2. It is placed into the lower lacrimal punctum immediately after PRK (bilaterally).
   3. The insert slowly dissolves over time.
2. Standard of care topical Fluorometholone (0.1% ophthalmic suspension) a. Tapered over time: i. 1 drop in each eye QID for 1 st week postop. ii. 1 drop in each eye TID for 2 nd week postop. iii. 1 drop in each eye BID for 3 rd week postop. iv. 1 drop in each eye qD for 4 th week postop. DURATION 1.Study subjects will be followed for 3 months after PRK. 2. Including recruitment, enrollment, treatment, and 3 months of follow-up, the study is expected to last 12 months total.

VISIT SCHEDULE

Subjects will be seen at 5 scheduled study visits (in addition to any unanticipated interim visits):

1. Preoperative
2. Operative
3. 1 week
4. 1 month
5. 3 months

NUMBER OF SUBJECTS Up to 60 subjects (120 eyes) will be enrolled to achieve the required treated eyes. Subjects will be treated with PRK bilaterally on one of the platforms (VISX, EX500, or equivalent) and will be randomized to receive one of two postoperative steroid regimens: Dextenza insert or standard of care topical Fluorometholone. DATA COLLECTION Data in this study will primarily be patient-generated. Investigators may also use patient health records, such as Genesis (e.g., for standard-of-care operative planning; verifying eligibility criteria). Investigators will prospectively collect data from eye examinations and questionnaires.

The schedule for standard of care eye testing and questionnaires (PROWL, COMTOL, and the Take Home questionnaire) is listed in Table 2, Section 10.2. Take Home questionnaires with a visual analogue scale and queries about postoperative medication use will be sent home with the patients to be completed postoperatively every day until the 1 Week visit. Prior to enrollment, clinic staff will flag patients who meet preoperative exam inclusion criteria and who agree to be referred to study investigators to obtain informed consent. Eligible subjects will sign Informed Consent and HIPAA Authorization forms. These forms include language permitting study investigators to use relevant data from a standard of care preoperative examination performed by clinic staff prior to the subject signing the Informed Consent and HIPAA Authorization forms. The purpose of using the previously gathered preoperative data is

To avoid a repeat preoperative visit, thus reducing patient and clinic burden and loss-to-follow- up. Preoperative and postoperative data will be added to the subject's study record and entered into an Excel Database.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 years of age and older, either active duty or dependents, who are eligible for care;
2. Myopia with manifest refractions ranging from 0.00 D to -8.00 D MRSE, with astigmatism ranging from 0.00 to -3.00 D CYL.
3. A stable refraction for the past year, as demonstrated by change in Sphere of ≤ 0.50 D and/or change in Cylinder of ≤ 0.50 D in the eyes to be treated;
4. A difference between cycloplegic and manifest refractions of

   ≤ 0.75 D MRSE in both eye(s);
5. BSCVA at least 20/20 in the treated eyes;
6. Discontinue use of contact lenses for at least 4 weeks (for hard lenses) or 2 weeks (for soft lenses) prior to the preoperative examination, and through entire study. The subject shall not be considered a contact lens wearer if they are not wearing hard contact lenses for 4 weeks or soft contact lenses for 2 weeks;
7. Central corneal thickness of at least 500 microns in the both eye(s);
8. Willing and able to return for scheduled follow-up examinations;
9. Able to provide written informed consent and follow study instructions in English.
10. Permission of the Commanding Officer for active duty subjects to receive refractive surgery and participate in the study.
11. Qualifies for treatment on all study lasers within FDA-approved parameters.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Postoperative Pain During the First Week Postoperative PRK | week 1 post surgery
  Assessed using a Take Home questionnaire for the first week postop that includes:
  * Visual analogue scale
  * Questions about medication utilization (adherence) and frequency
Self-Reported Intermediate-Term Postoperative Symptoms | pre-op, 1 week, 1 month, 3 month
  COMTOL questionnaire given to subjects at their pre and post operative visits
Epithelial Closure | 1 week, 1 month, 3 months
  Evaluated during post-op visits as yes/no. Evaluation will be done during the slit lamp examination
Incidence of Haze | Preop, post op 1 week, 1 month, 3 months
  Evaluated during the slit lamp examination and recorded as clinically significant haze Yes/no
Refractive Outcomes | pre-op, 1 week, 1 month, 3 months
  Measured in MRSE, Manifest Refraction and lines of vision loss

SECONDARY OUTCOMES:
Return to Duty | Pre-op, 1 week, 1 month, 3 months
  As measured by performance on the Combat Driving Simulator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee A, Blair HA. Dexamethasone Intracanalicular Insert: A Review in Treating Post-Surgical Ocular Pain and Inflammation. Drugs. 2020 Jul;80(11):1101-1108. doi: 10.1007/s40265-020-01344-6. PMID 32588339
- [Background] Brooks CC, Jabbehdari S, Gupta PK. Dexamethasone 0.4mg Sustained-Release Intracanalicular Insert in the Management of Ocular Inflammation and Pain Following Ophthalmic Surgery: Design, Development and Place in Therapy. Clin Ophthalmol. 2020 Jan 13;14:89-94. doi: 10.2147/OPTH.S238756. eCollection 2020. PMID 32021072
- [Background] Tyson SL, Campbell P, Biggins J, Driscoll A, Jarrett P, Gibson A, Vantipalli S, Metzinger JL, Goldstein MH. Punctum and canalicular anatomy for hydrogel-based intracanalicular insert technology. Ther Deliv. 2020 Mar;11(3):173-182. doi: 10.4155/tde-2020-0010. Epub 2020 Mar 16. PMID 32172659
- [Background] Cheng KJ, Hsieh CM, Nepali K, Liou JP. Ocular Disease Therapeutics: Design and Delivery of Drugs for Diseases of the Eye. J Med Chem. 2020 Oct 8;63(19):10533-10593. doi: 10.1021/acs.jmedchem.9b01033. Epub 2020 Jun 2. PMID 32482069
- [Background] McLaurin EB, Evans D, Repke CS, Sato MA, Gomes PJ, Reilly E, Blender N, Silva FQ, Vantipalli S, Metzinger JL, Gibson A, Goldstein MH. Phase 3 Randomized Study of Efficacy and Safety of a Dexamethasone Intracanalicular Insert in Patients With Allergic Conjunctivitis. Am J Ophthalmol. 2021 Sep;229:288-300. doi: 10.1016/j.ajo.2021.03.017. Epub 2021 Mar 25. PMID 33773984